CLINICAL TRIAL: NCT05213234
Title: Chronotherapy of 5-Aminosalicylic Acid in Ulcerative Colitis: A Randomized Crossover Trial
Brief Title: Chronotherapy of 5-Aminosalicylic Acid in Ulcerative Colitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ali Keshavarzian, Chief of the Section of Gastroenterology, Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20052807
Record Dates: First submitted 2021-12-09; First posted 2022-01-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Chronotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning Medication Administration (Other): Subjects are directed to take their medication between 06:00 and 10:00.
  Interventions: Behavioral: Chronotherapy
- Night Medication Administration (Other): Subjects are directed to take their medication between 18:00 and 22:00.
  Interventions: Behavioral: Chronotherapy

INTERVENTIONS:
Behavioral: Chronotherapy — Chronotherapy is a behavioral intervention that has the intended effect of maximizing therapeutic benefit of a drug by coordinating intake times and biological rhythms.

SUMMARY:
The hypothesis of this study is that appropriate time of day of administration of oral, once daily 5-ASA therapy in alignment with the host circadian rhythms will improve subclinical inflammation and microbial structure/function and increase mucosal 5-ASA levels.

All subjects will be randomized to once daily 5-ASA medications at two different times of the day: between 06:00 - 10:00 h or 18:00 - 22:00 h. Three disease assessments will performed at: 1) enrollment just before randomization; 2) month 3, at the completion of first arm (Condition 1), and 3) month 6, after completion of the second arm (Condition 2). During these study time points, participants will be asked to complete questionnaires, track their 5-ASA medication usage, provide a stool sample, blood draw, urine test, collect saliva, wear a watch to measure sleep patterns, and complete a flexible sigmoidoscopy.

ELIGIBILITY:
Inclusion Criteria: Study will include individuals that are;

1. M/F, 18-65 years of age
2. Ulcerative Colitis with Inactive Disease (Mayo Score ≤ 2; partial Mayo Score ≤ 1 with endoscopic score 0-1)
3. Subclinical inflammation stool calprotectin > 50 or CRP > mg/L above the upper limit of normal or PROMIS Fatigue Score ≥ 50)
4. Stable medications with no disease flares for the > 3 months,

Exclusion Criteria: Study will not include individuals that are;

1. Active UC at enrollment (Mayo > 2 and/or sigmoidoscopy score of 2 or 3)
2. Regular use of suppositories or enemas within the last 3 months ORA: 20052807-IRB01 Date IRB Approved: 11/6/2023 Amendment Date: 4/7/2024 Protocol Version Date: 4/4/2024 7
3. Use of biologics or immunomodulatory medications ( i.e. infliximab, Adalimumab, azathioprine, Vedolizumab, methotrexate, etc.)
4. Prior ostomy or subtotal colectomy
5. Recent prednisone or antibiotic use in last 12 weeks
6. Major Depression identified as Beck Depression Inventory (score ≥21)
7. Restless leg syndrome (score ≥ 15 on the IRLS Study Group Rating Scale)
8. Sleep apnea (score high risk ≥ 2 or more categories on the Berlin Questionnaire)
9. Clinically significant diabetes (Hgb-A1c>7)
10. Regular use of medications that affect intestinal permeability, intestinal motility and/or NSAIDs 4 weeks prior to the study
11. Clinically significant cardiac, renal (creatinine > twice normal) or liver disease
12. Alcohol use disorder (AUDIT>8)
13. Chronic use of illicit drugs
14. Shift Work
15. Inability to sign an informed consen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Stool Calprotectin from Baseline to Morning Medication Administration to Night Medication Administration | 10 minute stool collection at Baseline, 10 minute stool collection at Morning Medication Administration, and 10 minute stool collection at Night Medication Administration
  ELISA
Change in Mucosal 5-ASA Concentration from Baseline to Morning Medication Administration to Night Medication Administration | 30 minute flexible sigmoidoscopy at Baseline, 30 minute flexible sigmoidoscopy at Morning Medication Administration, and 30 minute flexible sigmoidoscopy at Night Medication Administration
  HPLC of tissue samples taken during flexible sigmoidoscopy at Baseline, Morning Medication Administration and Night Medication Administration

SECONDARY OUTCOMES:
Change in Intestinal Permeability from Baseline to Morning Medication Administration to Night Medication Administration | 24 hour urine collection at baseline, 24 hour urine collection at Morning Medication Administration, and 24 hour urine collection at Night Medication Administration
  Intestinal permeability is assessed through spectrophotometric measurements of sucralose, sucrose, maltose and lactulose concentrations in urine following ingestion of a sugar cocktail.
Change in Serum Cytokines from Baseline to Morning Medication Administration to Night Medication Administration | Single blood draw at baseline, single blood draw at Morning Medication Administration, and single blood draw at Night Medication Administration
  LBP, LPS, zonulin, and sCD14
Change in Mayo Score from Baseline to Morning Medication Administration to Night Medication Administration | 5 minute questionnaire at Baseline, 5 minute questionnaire at Morning Medication Administration, 5 minute questionnaire at Night Medication Administration
  Mayo Score
Change in Circadian Rhythms from Baseline to Morning Medication Administration to Night Medication Administration | Wrist Actigraphy Watch worn for two weeks at Baseline, two weeks at Morning Medication Administration, and two weeks at night medication administration
  Wrist Actigraphy

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - The Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No